CLINICAL TRIAL: NCT04430153
Title: Investigating the Actual Daily-life Upper Limb Activity Profile in Relation to Observed and Perceived Function in the Chronic Phase Post Stroke
Brief Title: What do I Think I Can do and What do I Really do: the Use of the Arm in Daily Life After Stroke
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Professor, KU Leuven
Other Study IDs: S64074; 1153320N (Other Grant/Funding Number: Research Foundation - Flanders (FWO))
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low match: A group with both low observed and perceived upper limb ability.
  Interventions: Other: "Class 1 Medical Device" CE certified devices: ActiGraph wGT3X-BT accelerometer
- Good match: A group with both good observed and perceived upper limb ability.
  Interventions: Other: "Class 1 Medical Device" CE certified devices: ActiGraph wGT3X-BT accelerometer
- Mismatch: A group with good observed but low perceived function.
  Interventions: Other: "Class 1 Medical Device" CE certified devices: ActiGraph wGT3X-BT accelerometer

INTERVENTIONS:
Other: "Class 1 Medical Device" CE certified devices: ActiGraph wGT3X-BT accelerometer — Accelerometers on both patients' wrists will give insight into the daily life upper limb use.

SUMMARY:
This study was organized to investigate the real upper limb use in persons after stroke. Persons after stroke often have problems moving their affected arm, leading to limitations in performing simple tasks. In previous research in a group of 60 patients post stroke the investigators investigated two things: they observed how patients can move their affected arm, and the investigators asked patients to indicate how they think they can use their affected arm. Surprisingly, the investigators concluded that in patients with a similar, good observed arm use there were two groups: (1) a 'match' group, reporting they can use their arm well, and (2) a 'mismatch' group, reporting they can not use their arm well. This project will further investigate this last group. The investigators will now use sensor technology to investigate the actual daily life arm use during daily life. The investigators hypothesize this daily arm use will be lower in the mismatch group than in the group with good observed and perceived ability.

DETAILED DESCRIPTION:
The investigators will perform a cross-sectional study to acquire insight into the actual daily-life UL activity profile of patients in the chronic phase post stroke. A sample of 60 community-dwelling patients more than six months after stroke will be recruited and will be investigated with both standardized clinical, patient-reported and sensor-based UL assessments. Our sample will include three groups of 20 patients with (1) both low observed and perceived function; (2) both good observed and perceived function; and (3) good observed but low perceived function, i.e. the mismatch group.

To better understand this mismatch group, it is pivotal to investigate daily arm and hand use in patients in the chronic phase after stroke as the investigators expect patients in the mismatch group to have significantly reduced arm and hand use throughout the day. After all, stroke rehabilitation interventions intend to improve patients' performance in daily life, but the objective evaluation of this aim is a challenge. Standardized assessments performed in the rehabilitation environment or patients' home do not validly reflect daily-life upper-limb use. To achieve insight into the observed upper limb function, apart from using internationally accepted observation-based assessments such as the FMA and SIS hand function, monitoring patients after stroke will also be performed using sensor-based systems.

The investigators hypothesize the mismatch group will show a comparable daily-life UL activity profile compared to patients with both low observed and perceived function. However, when compared to patients with good observed and perceived function, the mismatch group shows significantly reduced daily-life UL activity by means of sensor-based evaluation.

ELIGIBILITY:
Inclusion Criteria:

(1) unilateral, supratentorial stroke as defined by WHO; (2) minimum 6 months after stroke, and living in the community; (3) ≥ 18 years old; and (4) informed consent.

Exclusion Criteria:

(1) a musculoskeletal and/or other neurological disorder such as previous stroke, head injury, or Parkinson's disease that interfere with the protocol; and (2) severe communication or cognitive deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty patients with chronic stroke (>6 months post stroke) will be recruited
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer motor assessment - upper extremity | After inclusion
  Investigation of overall motor impairment of the affected upper limb: shoulder, arm, wrist, hand and fingers.
  Minimum: 0. Maximum: 66. Higher scores mean a better outcome.
Stroke Impact Scale 3.0 | After inclusion
  Self-reported outcome, measuring the impact of a stroke on activities, participation and quality of life, using the most affected body side.
  Minimum: 0. Maximum: 100, for each of the 9 domains assessed. Higher scores mean a better outcome.
Hours of use of each limb | After 3 days of sensor-based assessment
  Hours of use of each limb as measured with the accelerometer
Use ratio | After 3 days of sensor-based assessment
  Dividing hours of use of the affected limb by the hours of use of the non-affected limb
Magnitude ratio | After 3 days of sensor-based assessment
  The natural log of the vector magnitude of the non-dominant limb (or affected limb) divided by the vector magnitude of the dominant (or non-affected) limb
  The natural log of the vector magnitude of the non-dominant limb (or affected limb) divided by the vector magnitude of the dominant (or non-affected) limb Natural log of the vector magnitude of the affected divided by the non-affected limb
Bilateral magnitude | After 3 days of sensor-based assessment
  Sum of the vector magnitude from the two limbs

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | After inclusion
  Stroke severity. Minimum: 0. Maximum: 42. Higher scores mean worse outcome.
Modified Rankin Scale (mRS) | After inclusion
  Disability. Minimum: 0. Maximum: 42. Higher scores mean worse outcome. Minimum: 0. Maximum: 6. Higher scores mean worse outcome.
Montreal Cognitive Assessment (MoCA) | After inclusion
  Cognitive impairment. Minimum: 0. Maximum: 30. Higher scores mean better outcome.
Start Cancellation Test (SCT) | After inclusion
  Unilateral spatial neglect. Min: 0. Max: 54. Higher scores are better, scores <44 indicate the presence of USN.
Hospital Anxiety and Depression Scale (HADS) | After inclusion
  Anxiety and depression. Minimum: 0. Maximum: 42. Higher scores mean worse outcome.
Barthel Index (BI) | After inclusion
  Independence in activities of daily living. Minimum: 0. Maximum: 100. Higher scores mean better outcome.
Functional Ambulation Categories (FAC) | After inclusion
  Walking ability. Minimum: 0. Maximum: 5. Higher scores mean better outcome.
International Physical Activity Questionnaire (IPAQ) | After inclusion
  Patient-reported physical activity. 3 levels, higher levels are better.
Motor Activity Log Amount of Use (MAL AOU) - Dutch version | After inclusion
  Amount the individual uses the paretic arm. 26 items, per item: min. 0, max. 5. Higher scores mean better outcome.
ABILHAND | After inclusion
  Self-reported measure of (bi)manual ability in everyday activities. Rasch based logit scale. Higher logit scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No